CLINICAL TRIAL: NCT03321084
Title: Effects of MatPilates in Pain and Functionality in Elderly Woman With Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria das Graças Rodrigues de Araújo (Other)
Responsible Party: Sponsor-Investigator, Maria das Graças Rodrigues de Araújo, PhD, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MatPilates and Ostheoarthritis; Feedback N. 2.019.484 (Other: UFPE CAAE N. 63530416.1.0000.5208)
Record Dates: First submitted 2017-09-14; First posted 2017-10-25 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthrosis; Exercise Movement Techniques; Pilates; Elderly; Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Two groups: a MatPilates group (MG) and a Control group (CG).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The one who assess the patients in the beginning and in the final moment (investigator) not know in what group the patient is. As the investigator that will do the statistic (outcome assessor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MatPilates (Experimental): In the beginning was nominated Contrology, but today is known as Pilates. Created by Joseph Humbertus Pilates. This technique is based on respiration, balance, flexibility, proprioception and muscular strength. One of the main work is on the power house (core), biomechanical axis of the body, composed of muscles: rectus abdominis, paravertebral, multifidus, diaphragm, and those of the perineal center.
  Interventions: Other: MatPliates
- Control (Other): It continues in your daily life with phone monitoring.
  Interventions: Other: Control

INTERVENTIONS:
Other: MatPliates — The MatPilates program was specialized developed for this trial, in which all exercises belong to contemporaneous Pilates style. Each session has 60 minutes of duration, divided in three blocs (stretching, exercise and relaxation), with mean of 10, 40 and 10 minutes respectively (VIEIRA et al., 2016). Each exercise will be performed in one series of 10 to 15 repetitions and will be modified accordingly the patient need.
  Other Names: Experimental
  Arms: MatPilates
Other: Control — Will not be submitted to any physical intervention. It continues in your daily life with only phone monitoring.
  Arms: Control

SUMMARY:
Introduction: The osteoarthrosis is incurable, one of the most incapacitating disease around the world and your prevalence is increasing every year. The main consequences of this disease is pain and loss of functionality as a result of biomechanical limitations coming from articular inflammation. Among the variability of therapeutic resources, we propose MatPilates like a no drug intervention, that probably will contribute for a decrease in the symptoms of this disease.

Objective: It is hypothesized that MatPilates is a method capable of decrease pain and increase functionality in elderly woman with osteoarthrosis.

Methods: This study is a randomized double blind clinical trial, in which the volunteer need be in between 60 and 69 years old. Will be formed of two groups: MatPilates Group (MG) and Control Group (CG), and the ideal "n" will be calculated in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral osteoarthritis
* Body mass index (BMI) between 25 and 34,9 (WHO, 2000)
* Mini mental state examination score, with cutoff score of 18 (illiterate) and 24 (literate) (BRUCKI et al. 2003; LOURENÇO e VERAS, 2006)
* Unassisted gait (no wheelchair, no walking stick, no crutches or no walker)
* No history of neurologic disease
* No other physical activity
* Never practiced Pilates

Exclusion Criteria:

* Change in habitual drug's program during the study
* Join in other physical activity during the study
* Refuse to wear suitable clothing

Ages: 60 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
Pain. | 7 weeks.
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

SECONDARY OUTCOMES:
Pain | 7 weeks.
  Visual analog scale.
Pain | 7 weeks.
  Lequesne Index.
Functionality. | 7 weeks.
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
Functionality. | 7 weeks.
  Lequesne Index.
Stiffness. | 7 weeks.
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
Balance. | 7 weeks.
  Timed and Up Go Test (TUG)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Kinesiotherapy and Manual Therapeutic Resources, Department of Physical Therapy, Federal University of Pernambuco (UFPE), Recife, Pernambuco, Brazil